CLINICAL TRIAL: NCT01379482
Title: Phase II Study of Patients With Peritoneal Carcinomatosis From Gastric Cancer Treated With Preoperative Systemic Chemotherapy Followed by Peritonectomy and Intraperitoneal Chemotherapy
Brief Title: Neo-adjuvant Chemo + Peritonectomy + Hyperthermic Intraperitoneal Chemo in Peritoneal Carcinomatosis From Gastric Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Uppsala University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2007/073; 43145 (Other Grant/Funding Number: Uppsala University sådd-ALF)
Record Dates: First submitted 2011-06-07; First posted 2011-06-23 (Estimated); Last update posted 2014-05-06 (Estimated); Status verified 2011-05

CONDITIONS: Peritoneal Carcinomatosis; Gastric Cancer
Keywords: Peritoneal carcinomatosis from gastric cancer
MeSH Terms: conditions — Peritoneal Neoplasms; Stomach Neoplasms | interventions — Combined Modality Therapy; Fluorouracil; Paclitaxel

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Multimodal treatment (Experimental): Neoadjuvant systemic chemotherapy followed by cytoreductive surgery, hyperthermic intraperitoneal chemotherapy and early postoperative intraperitoneal chemotherapy
  Interventions: Drug: Multimodal treatment

INTERVENTIONS:
Drug: Multimodal treatment — 3 months (range 2-4.5) with neoadjuvant systemic chemotherapy. Four weeks after receiving the last course of chemotherapy, patients will undergo laparotomy with the objective of performing cytoreduction + hyperthermic intraperitoneal chemotherapy.
  Early peritoneal chemotherapy though intrabdominal drains for the first five postoperative days.
  Neo-adjuvant chemotherapy:
  Irinotecan+Nordic FLv (6 pat.) EOX (6 pat.) FLOX (3 pat.) Docetaxel+Irinotecan+5-FU+LV (1 pat.) FOLFIRI (1 pat.) ECF (1 pat.)
  Hyperthermic intraoperative chemotherapy:
  Cisplatin+doxorubicin (5 pat.). Oxaliplatin +concomitant i.v. 5-FU+ i.v. LV (3 pat.)
  Early postoperative chemotherapy:
  5-FU + i.v. LV (5 pat.) Paclitaxel (1 pat.)
  Other Names: Irinotecan+Nordic FLv (6 pat.); EOX (6 pat.); FLOX (3 pat.); Docetaxel+Irinotecan+5-FU+LV (1 pat.); FOLFIRI (1 pat.); ECF (1 pat.); Cisplatin+doxorubicin (5 pat.).; Oxaliplatin +concomitant i.v. 5-FU+ i.v. LV (3 pat.); 5-FU + i.v. LV (5 pat.); Paclitaxel (1 pat.)

SUMMARY:
The aims of this study are to investigate whether multimodal treatment of peritoneal carcinomatosis from gastric cancer is feasible and to evaluate the clinical outcomes and clinical effectiveness of neoadjuvant systemic chemotherapy followed by cytoreductive surgery + hyperthermic intraperitoneal chemotherapy + early postoperative intraperitoneal chemotherapy, as compared to systemic chemotherapy only, in patients with peritoneal carcinomatosis from gastric cancer.

DETAILED DESCRIPTION:
Between January 2005 and March 2009, 18 consecutive patients with PC from gastric cancer were scheduled for neoadjuvant systemic chemotherapy followed by CRS+HIPEC+EPIC at Uppsala University Hospital, Uppsala, Sweden. The regional ethics committee approved the study and informed consent was obtained from each patient and the study was registered in ClinicalTrials.gov, with identifier NCT01379482. The eligibility requirements for treatment were: histologically confirmed diagnosis of primary gastric adenocarcinoma; histologically and radiologically confirmed PC diagnosis; no distant metastases; adequate renal, haematopoietic and liver functions, and Karnofsky performance status (KPS) of > 70. Table 1 summarises demographic and basic clinical patient data.

Patients Eighteen patients (eight female and ten male), with a median age of 57 years (range 38-74), were included in the study. Treatment began with three months' (range 2-4.5) neoadjuvant systemic chemotherapy. Four weeks after receiving the last course of chemotherapy, patients with no clinical and radiological signs of tumour progression underwent laparotomy in preparation for CRS+HIPEC followed by EPIC for five days. Patients with clinical and radiological signs of tumour progression during the neoadjuvant systemic chemotherapy did not undergo the planned loco-regional treatment but continued with palliative systemic chemotherapy at the discretion of the physician in charge of the patient.

Neoadjuvant chemotherapy The intention was to treat the patients with combination chemotherapy for three months. The choice of chemotherapy was individualised, but all patients received optimal drug combinations suitable for good performance patients with metastatic gastric cancer.

Routine clinical controls and blood sampling were done before every treatment cycle. In order to rule out patients with progressive disease and distant metastasis, abdominal and thoracic CT scan evaluations were performed prior to surgery.

Surgical treatment Depending on disease extent, CRS was performed as described by Sugarbaker. Immediately postoperatively, tumour load and completeness of cytoreduction for PC were recorded using the Peritoneal Cancer Index (PCI) [12] and Completeness of Cytoreduction scores (CC) respectively. The PCI (range 1-39) consists of lesion size scores in 13 different regions of the abdomen: 0=no tumour seen, 1=tumour up to 0.5 cm, 2=tumour up to 5 cm and 3=tumour>5 cm. The PCI score is calculated by adding together the lesion size scores for the 13 regions. The CC score is based upon the size of tumour left after cytoreduction: CC0=no peritoneal seeding visible, CC1=nodules up to 2.5 mm, CC2=nodules up to 2.5 cm and CC3=nodules>2.5 cm.

HIPEC and EPIC HIPEC was administered according to the Coliseum technique and was combined with EPIC for five days. Before perfusion, the patient's body temperature was lowered to 35°C with a cooling blanket (Allon®). The intra-abdominal temperature during perfusion ranged from 42°C to 44°C. Four intra-abdominal drains were left in place after surgery and EPIC was given daily during the first five postoperative days.

Tumour markers, histopathology and adverse events Five serum tumour markers (CEA, CA 125, CA 19-9, CA 15-3 and CA 72-4) were taken one to six days before surgery and ten days after surgery, to analyse the frequency of the impact of gastric cancer with PC on these tumour markers.

The sixth edition of the TNM classification was used. The presence of signet ring cells and the grade of differentiation according to Lauren's classification were reported.

Therapy-related adverse events were graded according to the National Cancer Institute's common toxicity criteria (NCI-CTC) version 3.0. OS was calculated for all patients from the date of the first neoadjuvant chemotherapy.

Statistical methods All analyses were performed on the basis of intention-to-treat. OS and disease-free survival (DFS) were analysed for patients treated with CC0. Results were presented as the median, with a 95% confidence interval (CI). A P-value of less than 0.05 was considered statistically significant. The computer software package STATISTICA AXA version 10.0, StatSoft Scandinavia, Sweden, was used for statistical evaluation of the survival data.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed diagnosis of primary gastric cancer + histologically and/or radiologically confirmed peritoneal carcinomatosis diagnosis
* Adequate renal-, hematopoietic- and liver functions
* WHO performance status (WHO) of < 2.

Exclusion Criteria:

* Distant metastases
* Surgically not resectable lymph-node metastasis
* Contraindication to chemotherapy treatment

Max Age: 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2005-01; Primary Completion 2009-03 (Actual); Study Completion 2009-03 (Actual)

PRIMARY OUTCOMES:
Overall survival | Jan 2005 until Mars 2009

CONTACTS AND LOCATIONS:
Overall Officials: Haile Mahteme, Ass prof, Principal Investigator — Uppsala University, Sweden
Locations (1):
- Uppsala University, Uppsala, Sweden